CLINICAL TRIAL: NCT01611090
Title: Randomized, Double-blind, Placebo-controlled Phase 3 Study of Ibrutinib, a Bruton's Tyrosine Kinase (BTK) Inhibitor, in Combination With Bendamustine and Rituximab (BR) in Subjects With Relapsed or Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: A Study of Ibrutinib in Combination With Bendamustine and Rituximab in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR100840; PCI-32765CLL3001 (Other: Janssen Research & Development, LLC); 2012-000600-15 (EudraCT Number); U1111-1135-3745 (Other: Universal Trial Number)
Record Dates: First submitted 2012-05-15; First posted 2012-06-04 (Estimated); Results first posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: Chronic lymphocytic leukemia; Small lymphocytic lymphoma; Relapsed or refractory chronic lymphocytic leukemia; Relapsed or refractory small lymphocytic lymphoma; Ibrutinib; PCI-32765; JNJ-54179060; Bruton's tyrosine kinase inhibitor; Bendamustine; Rituximab
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence | interventions — ibrutinib; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ibrutinib + BR (Experimental): Ibrutinib 420 mg will be administered orally once daily on a continuous schedule. All subjects will receive background therapy with bendamustine and rituximab (BR) for a maximum of 6 cycles (a cycle is defined as 28 days, with the exception of Cycle 1, which will be 29 days to allow for rituximab dosing prior to bendamustine and study medication).
  Interventions: Drug: Ibrutinib; Drug: Bendamustine hydrochloride; Drug: Rituximab
- Placebo + BR (Placebo Comparator): Matching placebo will be administered orally once daily on a continuous schedule. All subjects will receive background therapy with BR for a maximum of 6 cycles (a cycle is defined as 28 days, with the exception of Cycle 1, which will be 29 days to allow for rituximab dosing prior to bendamustine and study medication).
  Interventions: Drug: Bendamustine hydrochloride; Drug: Rituximab; Drug: Placebo

INTERVENTIONS:
Drug: Ibrutinib — Type=exact number, unit=mg, number=420 , form=capsule, route=oral use. Capsule is taken once daily continuously.
  Arms: Ibrutinib + BR
Drug: Bendamustine hydrochloride — Type=exact number, unit=mg, number=70 mg/m2, route=intravenous use. Administered intravenously on Cycle 1, Days 2-3 and Cycles 2-6, Days 1-2.
Drug: Rituximab — Type=exact number, unit=mg, number=375 mg/m2 and 500 mg/m2, route=intravenous use. Administered intravenously on Cycle 1, Day 1, and Cycles 2-6, Day 1, respectively.
Drug: Placebo — Form=capsule, route=oral use. Capsule is taken once daily continuously.
  Arms: Placebo + BR

SUMMARY:
The purpose of this study is to examine the safety and efficacy of Ibrutinib administered in combination with bendamustine and rituximab in patients with relapsed or refractory chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL).

DETAILED DESCRIPTION:
This is a randomized (patients will be assigned by chance to study treatments), double-blind (patients and study personnel will not know the identity of study treatments), placebo (an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial)-controlled study to determine the benefits and risks of combining ibrutinib with bendamustine and rituximab (BR) in patients with relapsed or refractory CLL/SLL following at least 1 line of prior systemic therapy. Approximately 580 patients will be randomized in a 1:1 ratio to either treatment arm A (placebo) or treatment arm B (ibrutinib 420 mg).

Study medication will be administered orally once daily on a continuous schedule. All patients will receive BR as the background therapy plus either ibrutinib or placebo for a maximum of 6 cycles, after which treatment with ibrutinib or placebo will continue until disease progression or unacceptable toxicity.

A treatment cycle will be defined as 28 days. The study will include a screening phase, a treatment phase, and a follow-up phase. Study end is defined as when either 80% of the patients have died or 5 years after the last patient is randomized into the study, whichever occurs first.

Patients in treatment arm A (placebo) who complete the treatment phase, with disease progression or (after interim analysis) meet International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria for treatment, may crossover to ibrutinib treatment (as in treatment arm B), at the investigators discretion. This open-label, next-line treatment with ibrutinib will continue until disease progression, unacceptable toxicity, withdrawal from study, or until the study end, whichever occurs earlier. One interim analysis is planned for the study. Efficacy evaluations will include computed tomography scans, laboratory testing, focused physical examinations, bone marrow biopsy and aspirate, and assessment of patient-reported outcomes. In both treatment arms, samples for the development of a population-based pharmacokinetic (PK; study of what the body does to a drug) approach will be collected. Safety will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) that meets protocol-defined criteria
* Active disease meeting at least 1 of the International Workshop on Chronic Lymphocytic Leukemia 2008 criteria for requiring treatment
* Measurable nodal disease by computed tomography
* Relapsed or refractory CLL or SLL following at least 1 prior line of systemic therapy consisting of at least 2 cycles of a chemotherapy-containing regimen
* Eastern Cooperative Oncology Group Performance Status score of 0 or 1
* Hematology and biochemical values within protocol-defined limits
* Agrees to protocol-defined use of effective contraception
* Women of childbearing potential must have negative blood or urine pregnancy test at screening

Exclusion Criteria:

* Recent therapeutic interventions within 3 (chemotherapy/radiotherapy) to 10 weeks (immunotherapy)
* Prior treatment with ibrutinib or other Bruton's tyrosine kinase inhibitors or prior randomization in any other clinical study evaluating ibrutinib
* The presence of deletion of the short arm of chromosome 17
* Patients previously treated with a bendamustine-containing regimen who did not achieve a response or who relapsed and required treatment within 24 months of treatment with that regimen
* Patients for whom the goal of therapy is tumor debulking prior to stem cell transplant
* Received a hematopoietic stem cell transplant
* Known central nervous system leukemia/lymphoma or Richter's transformation
* Patients with uncontrolled autoimmune hemolytic anemia or autoimmune thrombocytopenia
* Chronic use of corticosteroids
* History of prior malignancy, except: malignancy treated with curative intent and with no known active disease present for >=3 years before randomization; adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease; adequately treated cervical carcinoma in situ without evidence of disease
* History of stroke or intracranial hemorrhage within 6 months prior to randomization; or clinically significant cardiovascular disease
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists or treatment with strong CYP3A4/5 inhibitors
* Known history of human immunodeficiency virus or hepatitis C, or active infection with hepatitis B or C
* Any uncontrolled active systemic infection or any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the patient's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk
* A woman who is pregnant or breast feeding, or a man who plans to father a child while enrolled in this study or within 3 months after the last dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 578 (Actual)
Dates: Start 2012-09-19 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (155):
- United States (42):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Berkeley, California
  - Duarte, California
  - Greenbrae, California
  - Stamford, Connecticut
  - Washington D.C., District of Columbia
  - Boca Raton, Florida
  - Jacksonville, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Chicago, Illinois
  - Springfield, Illinois
  - Fort Wayne, Indiana
  - Goshen, Indiana
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Westwood, Kansas
  - Louisville, Kentucky
  - Paducah, Kentucky
  - Marrero, Louisiana
  - Baltimore, Maryland
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Battle Creek, Michigan
  - Detroit, Michigan
  - Lansing, Michigan
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Lebanon, New Hampshire
  - Hackensack, New Jersey
  - Albuquerque, New Mexico
  - Dunkirk, New York
  - Hawthorne, New York
  - New York, New York
  - Bismarck, North Dakota
  - Cleveland, Ohio
  - Portland, Oregon
  - Charleston, South Carolina
  - Sioux Falls, South Dakota
  - Temple, Texas
  - Morgantown, West Virginia
- Argentina (3):
  - Buenos Aires
  - Ciudad Autonoma Buenos Aires
  - Córdoba
- Belgium (5):
  - Aalst
  - Bruges
  - Brussels
  - Ghent
  - Leuven
- Brazil (3):
  - Rio de Janeiro
  - Salvador
  - São Paulo
- Canada (7):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Hamilton, Ontario
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Colombia (2):
  - Bogotá
  - Floridablanca
- Czechia (2):
  - Brno
  - Prague
- France (7):
  - Créteil
  - Montpellier
  - Paris
  - Pessac
  - Pierre-Bénite
  - Tours
  - Villejuif
- Germany (22):
  - Aschaffenburg
  - Augsburg
  - Cologne
  - Dresden
  - Erlangen
  - Essen
  - Frankfurt
  - Frechen
  - Hamm
  - Heidelberg
  - Homburg/Saar
  - Kassel
  - Kiel
  - Koblenz
  - Kÿln N/a
  - Lebach
  - Magdeburg
  - Mannheim
  - Marburg
  - Mutlangen
  - Ulm
  - Würzburg
- Greece (2):
  - Athens
  - Thessalonikis
- Israel (7):
  - Haifa
  - Jerusalem
  - Nahariya
  - Netanya
  - Petah Tikva
  - Ramat Gan
  - Tel Aviv
- Mexico (3):
  - México
  - Monterrey
  - Oaxaca City
- Poland (5):
  - Brzozów
  - Chorzów
  - Krakow
  - Opole
  - Słupsk
- Portugal (4):
  - Coimbra
  - Lisbon
  - Ponta Delgada
  - Porto
- Russia (14):
  - Arkhangelsk
  - Dzerzhinsk
  - Krasnodar
  - Moscow
  - Nizhny Novgorod
  - Obninsk
  - Perm
  - Rostov-on-Don
  - Ryazan
  - Saint Petersburg
  - Samara
  - Sochi
  - Syktyvkar
  - Yekaterinburg
- Seoul, South Korea
- Spain (5):
  - Barcelona
  - L'Hospitalet de Llobregat
  - Madrid
  - Salamanca
  - Valencia
- Sweden (4):
  - Gothenburg
  - Huddinge
  - Stockholm
  - Umeå
- Turkey (Türkiye) (4):
  - Ankara
  - Istanbul
  - Izmir
  - Kayseri
- Ukraine (8):
  - Cherkassy
  - Dnipro
  - Donetsk
  - Khakhiv
  - Khmelnitskiy
  - Kiev
  - Lviv
  - Vinnitsa
- United Kingdom (5):
  - Birmingham
  - Harrow
  - Plymouth
  - Sheffield Yorks
  - Sutton

REFERENCES:
- [Derived] Abuhelwa AY, Almansour SA, Brown JR, Al-Shamsi HO, Abuhelwa Z, Kharaba Z, Bustanji Y, Semreen MH, Ali S, Alhuraiji A, McKinnon RA, Sorich MJ, Alzoubi KH, Hopkins AM. Statin use and survival in CLL/SLL treated with ibrutinib: pooled analysis of 4 randomized controlled trials. Blood Adv. 2025 Jul 22;9(14):3566-3575. doi: 10.1182/bloodadvances.2024015287. PMID 40266025
- [Derived] Fraser GAM, Chanan-Khan A, Demirkan F, Santucci Silva R, Grosicki S, Janssens A, Mayer J, Bartlett NL, Dilhuydy MS, Loscertales J, Avigdor A, Rule S, Samoilova O, Pavlovsky MA, Goy A, Mato A, Hallek M, Salman M, Tamegnon M, Sun S, Connor A, Nottage K, Schuier N, Balasubramanian S, Howes A, Cramer P. Final 5-year findings from the phase 3 HELIOS study of ibrutinib plus bendamustine and rituximab in patients with relapsed/refractory chronic lymphocytic leukemia/small lymphocytic lymphoma. Leuk Lymphoma. 2020 Dec;61(13):3188-3197. doi: 10.1080/10428194.2020.1795159. Epub 2020 Aug 6. PMID 32762271
- [Derived] Lavezzi SM, de Jong J, Neyens M, Cramer P, Demirkan F, Fraser G, Bartlett N, Dilhuydy MS, Loscertales J, Avigdor A, Rule S, Samoilova O, Goy A, Ganguly S, Salman M, Howes A, Mahler M, De Nicolao G, Poggesi I. Systemic Exposure of Rituximab Increased by Ibrutinib: Pharmacokinetic Results and Modeling Based on the HELIOS Trial. Pharm Res. 2019 May 1;36(7):93. doi: 10.1007/s11095-019-2605-8. PMID 31044267
- [Derived] Brown JR, Moslehi J, O'Brien S, Ghia P, Hillmen P, Cymbalista F, Shanafelt TD, Fraser G, Rule S, Kipps TJ, Coutre S, Dilhuydy MS, Cramer P, Tedeschi A, Jaeger U, Dreyling M, Byrd JC, Howes A, Todd M, Vermeulen J, James DF, Clow F, Styles L, Valentino R, Wildgust M, Mahler M, Burger JA. Characterization of atrial fibrillation adverse events reported in ibrutinib randomized controlled registration trials. Haematologica. 2017 Oct;102(10):1796-1805. doi: 10.3324/haematol.2017.171041. Epub 2017 Jul 27. PMID 28751558
- [Derived] Chanan-Khan A, Cramer P, Demirkan F, Fraser G, Silva RS, Grosicki S, Pristupa A, Janssens A, Mayer J, Bartlett NL, Dilhuydy MS, Pylypenko H, Loscertales J, Avigdor A, Rule S, Villa D, Samoilova O, Panagiotidis P, Goy A, Mato A, Pavlovsky MA, Karlsson C, Mahler M, Salman M, Sun S, Phelps C, Balasubramanian S, Howes A, Hallek M; HELIOS investigators. Ibrutinib combined with bendamustine and rituximab compared with placebo, bendamustine, and rituximab for previously treated chronic lymphocytic leukaemia or small lymphocytic lymphoma (HELIOS): a randomised, double-blind, phase 3 study. Lancet Oncol. 2016 Feb;17(2):200-211. doi: 10.1016/S1470-2045(15)00465-9. Epub 2015 Dec 5. PMID 26655421

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 578 participants were enrolled in the study. Among these, 289 participants were randomized in each ibrutinib + bendamustine/rituximab (BR) treatment group and placebo+BR treatment group.
Groups:
- Ibrutinib+BR: Participants received ibrutinib 420 milligram (mg) (3 * 140 mg capsules) orally once daily starting on Cycle 1 Day 2 for a maximum of 6 cycles (each cycle of 28 days except Cycle 1 which was of 29 days) along with BR. After 6 cycles ibrutinib alone was administered until disease progression or unacceptable toxicity.
- Placebo+BR: Participants received placebo (3 capsules) orally once daily starting on Cycle 1 Day 2 for a maximum of 6 cycles (each cycle of 28 days except Cycle 1 which was of 29 days) along with BR. After 6 cycles placebo alone was administered until disease progression or unacceptable toxicity.
- Crossover to Ibrutinib: Participants in the placebo+BR treatment group could cross over to receive next-line ibrutinib treatment (420 mg [3 * 140 mg capsules] orally once daily on a 28-day cycle) at the discretion of the investigator at the time of disease progression or if International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria for treatment were met.
Period: Randomized Period
Arm/Group | Ibrutinib+BR | Placebo+BR | Crossover to Ibrutinib
Started | 289 | 289 | 0
Treated | 287 | 287 | 0
Completed | 259 | 260 | 0
Not Completed | 30 | 29 | 0
Not completed — Lost to Follow-up | 8 | 3 | 0
Not completed — Withdrawal by Subject | 22 | 26 | 0
Period: Cross Over (Placebo to Ibrutinib)
Arm/Group | Ibrutinib+BR | Placebo+BR | Crossover to Ibrutinib
Started | 0 | 0 | 183
Treated | 0 | 0 | 183
Completed | 0 | 0 | 178
Not Completed | 0 | 0 | 5
Not completed — Lost to Follow-up | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibrutinib+BR | Placebo+BR | Total
Number analyzed (Participants) | 289 | 289 | 578
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (9.82) | 63.3 (9.3) | 63.5 (9.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 100 | 196
  Male | 193 | 189 | 382
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 21 | 34
  Not Hispanic or Latino | 256 | 253 | 509
  Unknown or Not Reported | 20 | 15 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 264 | 264 | 528
  Black | 8 | 6 | 14
  Asian | 1 | 2 | 3
  American Indian or Alaska Native | 1 | 1 | 2
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  Other | 3 | 7 | 10
  Unknown or not reported | 12 | 9 | 21
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 3 | 3 | 6
  BELGIUM | 14 | 14 | 28
  BRAZIL | 10 | 12 | 22
  CANADA | 27 | 35 | 62
  COLOMBIA | 0 | 1 | 1
  CZECH REPUBLIC | 12 | 11 | 23
  FRANCE | 16 | 11 | 27
  GERMANY | 10 | 11 | 21
  GREECE | 12 | 5 | 17
  ISRAEL | 14 | 12 | 26
  MEXICO | 1 | 2 | 3
  POLAND | 19 | 20 | 39
  PORTUGAL | 7 | 12 | 19
  RUSSIAN FEDERATION | 50 | 50 | 100
  SOUTH KOREA | 0 | 1 | 1
  SPAIN | 9 | 9 | 18
  SWEDEN | 2 | 4 | 6
  TURKEY | 24 | 27 | 51
  UKRAINE | 16 | 14 | 30
  UNITED KINGDOM | 5 | 9 | 14
  UNITED STATES | 38 | 26 | 64

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the interval between the date of randomization and the date of disease progression or death, whichever was first reported. IWCLL 2008 criteria for PD: New enlarged nodes >1.5 cm, new hepatomegaly or splenomegaly, or other new organ infiltrates, bone lesion, ascites, or pleural effusion confirmed due to chronic lymphocytic leukemia (CLL); >=50% increase in existing lymph nodes; >=50% increase in enlargement of liver or spleen; >=50% increase from baseline in lymphocyte count (and to >=5*10^9/L) or >=50% increase from nadir count confirmed on >=2 serial assessments if absolute lymphocyte count (ALC) >=30,000 per microliter and lymphocyte doubling time is rapid, unless considered treatment-related lymphocytosis; new cytopenia (Hemoglobin b [Hgb] or platelets) attributable to CLL; and transformation to a more aggressive histology.
Time Frame: Up to 5 years
Population: Intent to treat (ITT) population included all participants randomized into the study regardless of treatment actually received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ibrutinib+BR | Placebo+BR
Number analyzed (Participants) | 289 | 289
Months | 65.12 [55.43 to NA] — Here, NA indicates upper limit of confidence interval (CI) was not estimable due to insufficient number of events. | 14.32 [13.86 to 16.62]
Statistical Analysis 1: Comparison: Ibrutinib+BR vs Placebo+BR; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.229, 95% CI 2-sided [0.183 to 0.286]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR defined as number of participants achieving a complete response (CR), complete response with incomplete marrow recovery (CRi), nodular partial response (nPR) or partial response (PR). IWCLL 2008 criteria: CR- No lymphadenopathy and hepatosplenomegaly, no constitutional symptoms, neutrophils >1.5*10^9/liter (L), platelets >100*10^9/L, Hgb >11 gram per deciliter (g/dL) and absolute lymphocyte count <4000/microliter (mcL); CRi- CR with incomplete recovery of bone marrow; nPR- participants meet criteria for CR, but the bone marrow biopsy shows B-lymphoid nodules, may represent a clonal infiltrate; PR-2 of the following when abnormal at baseline: >=50% decrease in ALC, >=50% decrease in sum products of up to 6 lymph nodes, >=50% decrease in enlargement of spleen or liver; and 1 of the following: neutrophils >1.5*10^9/L, Platelets >100*10^9/L and Hgb>11 g/dL or >=50% improvement over baseline in any of these; no new enlarged nodes or new hepatosplenomegaly.
Time Frame: Up to 5 years
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ibrutinib+BR | Placebo+BR
Number analyzed (Participants) | 289 | 289
Percentage of participants | 87.2 | 66.1

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the interval between the date of randomization and the date of death from any cause.
Time Frame: Up to 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ibrutinib+BR | Placebo+BR
Number analyzed (Participants) | 289 | 289
Months | NA [70.93 to NA] — Here, NA indicates median and upper limit of CI was not estimable due to insufficient number of events. | NA [NA to NA] — Here, NA indicates median and CI was not estimable due to insufficient number of events.

4. Secondary Outcome: Percentage of Participants With Minimal Residual Disease (MRD)-Negative Response
Description: MRD-negative response was defined as the percentage of participants who reach MRD negative disease status (less than 1 chronic lymphocytic leukemia [CLL] cell per 10,000 leukocytes) in either bone marrow or peripheral blood. All randomized participants were included in this analysis. Participants with missing MRD data were considered non-responders.
Time Frame: Up to 5 years
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ibrutinib+BR | Placebo+BR
Number analyzed (Participants) | 289 | 289
Percentage of participants | 28.7 | 5.9

5. Secondary Outcome: Percentage of Participants With Sustained Hematologic Improvement
Description: Sustained hematologic improvement was defined as hematological improvement that was sustained continuously for greater than or equal to (>=) 56 days without blood transfusion or growth factors: 1) Platelet counts greater than (>)100* 109/liter (L) if baseline less than or equal to (<=) 100*109/L or increase >= 50 percent (%) over baseline; 2) Hemoglobin >11 gram per deciliters (g/dL) if baseline <= 11 g/dL or increase >= 2 g/dL over baseline.
Time Frame: Up to 5 years
Population: ITT population included all participants randomized into the study regardless of treatment actually received.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ibrutinib+BR | Placebo+BR
Number analyzed (Participants) | 289 | 289
Percentage of Participants
  Hemoglobin | 36.7 | 29.1
  Platelets | 30.8 | 21.8

6. Secondary Outcome: Median Time to Clinically Meaningful Improvement in FACIT-Fatigue Scale
Description: Time to improvement is defined as the time interval (months) from randomization to the first observation of improvement. FACIT-Fatigue is an instrument for use as a measure of the effect of fatigue in patients with cancer and other chronic diseases. Responses to the 13-item FACIT Fatigue Scale are reported on a 5-point categorical response scale ranging from 0 (not at all) to 4 (very much). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worst score) to 52 (best score).
Time Frame: Up to 2 years
Population: ITT population included all participants randomized into the study regardless of treatment actually received.
Measure: Number (95% Confidence Interval); unit: Months
Arm/Group | Ibrutinib+BR | Placebo+BR
Number analyzed (Participants) | 289 | 289
Months | 6.5 [4.7 to 10.7] | 4.6 [2.8 to 6.4]

7. Secondary Outcome: Number of Participants With Clinically Relevant Shifts in Disease-Related Symptoms
Description: The disease-related symptoms included fatigue, weight loss, fevers, night sweats, abdominal discomfort/splenomegaly and anorexia.
Time Frame: From the date of randomization to disease progression (Up to 2 years)
Population: ITT population included all participants randomized into the study regardless of treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib+BR | Placebo+BR
Number analyzed (Participants) | 289 | 289
Participants | 0 | 0

8. Secondary Outcome: Number of Participants Who Received Subsequent Antineoplastic Therapy
Description: Number of participants who received subsequent antineoplastic therapy was reported.
Time Frame: Up to 5 years
Population: Safety analysis set included all the randomized participants who received at least 1 dose of study drug or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib+BR | Placebo+BR
Number analyzed (Participants) | 287 | 287
Participants | 52 | 61

9. Secondary Outcome: Change From Baseline in Beta2 Microglobulin at End of Treatment (EOT)
Description: Change from baseline in beta2 microglobulin at end of treatment at time of primary analysis was reported.
Time Frame: Baseline to EOT (Up to 2 years)
Population: ITT population included all participants randomized into the study regardless of treatment actually received. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this endpoint.
Measure: Mean (Standard Deviation); unit: milligram per liter (mg/L)
Arm/Group | Ibrutinib+BR | Placebo+BR
Number analyzed (Participants) | 39 | 106
milligram per liter (mg/L) | -0.46 (1.77) | -0.23 (2.08)

10. Secondary Outcome: Change From Baseline in FACIT-Fatigue Scale at End of Treatment
Description: FACIT-Fatigue is an instrument for use as a measure of the effect of fatigue in patients with cancer and other chronic diseases. Responses to the 13-item FACIT Fatigue Scale are reported on a 5-point categorical response scale ranging from 0 (not at all) to 4 (very much). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worst score) to 52 (best score).
Time Frame: Baseline to EOT (up to 2 years)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ibrutinib+BR | Placebo+BR
Number analyzed (Participants) | 38 | 104
Units on a scale | -0.9 (11.22) | 0.0 (11.01)

11. Secondary Outcome: Change From Baseline in EORTC QLQ-C30 Physical Functioning Score at End of Treatment
Description: EORTC QLQ-C30 Physical Functioning Score is a questionnaire to assess quality of life of cancer patients. It is composed of 30 items, multi-item measure (28 items) and 2 single-item measures. For the multiple item measure, 4-point scale is used and the score for each item range from "1 = not at all" to "4 = very much". Higher scores indicate worsening. The 2 single-item measure involves question about the overall health and overall quality of life which was rated on a 7-point scale ranging from "1 = very poor" to "7 = excellent". Lower scores indicate worsening. All scale and item scores were linearly transformed to be in range from 0-100. A higher score represents a higher (better) level of functioning, or a higher (worse) level of symptoms.
Time Frame: Baseline to EOT (up to 2 years)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ibrutinib+BR | Placebo+BR
Number analyzed (Participants) | 38 | 104
Units on a scale | -2.1 (16.34) | -4.1 (22.52)

12. Secondary Outcome: Change From Baseline in EORTC QLQ-CLL 16 Domain Scores at End of Treatment
Description: The EORTC QLQ-CLL 16 is a 16-item disease specific module that comprises 5 domains of patient-reported health status important in CLL. There are three multi-item scales that include fatigue (2 items), treatment side effects and disease symptoms (8 items), and infection (4 items), and 2 single-item scales on social activities and future health worries. Responses are measured on a 4 point scale ranging from 1 (not at all) to 4 (very much).
Time Frame: Baseline to EOT (up to 2 years)
Population: ITT population included all participants randomized into the study regardless of treatment actually received. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this endpoint. Here, 'n' signifies the number of participants analyzed for the specified symptoms.
Measure: Mean (Standard Deviation); unit: Units on the scale
Arm/Group | Ibrutinib+BR | Placebo+BR
Number analyzed (Participants) | 38 | 104
Units on the scale
  Lost weight | 0.1 (0.86) | 0.0 (0.74)
  Dry mouth | 0.3 (0.96) | 0.1 (0.85)
  Bruises | 0.1 (0.61) | 0.0 (0.65)
  Abdominal discomfort: number analyzed (Participants) | 37 | 104
  Abdominal discomfort | 0.1 (0.81) | 0.0 (0.76)
  Temperature going up and down | 0.1 (0.93) | 0.0 (0.72)
  Night sweats: number analyzed (Participants) | 38 | 103
  Night sweats | -0.6 (0.92) | -0.3 (1.07)
  Skin problems: number analyzed (Participants) | 37 | 104
  Skin problems | 0.4 (1.14) | 0.3 (0.96)
  Feel ill | 0.1 (1.08) | 0.2 (0.98)
  Feel lethargic | 0.1 (1.01) | 0.0 (0.91)
  Felt slowed down: number analyzed (Participants) | 38 | 103
  Felt slowed down | 0.3 (0.80) | 0.0 (0.97)
  Limited in planning activities: number analyzed (Participants) | 38 | 103
  Limited in planning activities | 0.2 (0.97) | 0.1 (0.90)
  Worried about health in the future: number analyzed (Participants) | 38 | 103
  Worried about health in the future | 0.0 (0.94) | 0.0 (0.97)
  Trouble with chest infections | 0.2 (1.05) | 0.0 (0.82)
  Trouble with other infections | 0.7 (1.07) | 0.1 (0.86)
  Repeated courses of antibiotics | 0.9 (1.22) | 0.0 (0.97)
  Worried about picking up infection: number analyzed (Participants) | 38 | 103
  Worried about picking up infection | 0.3 (0.96) | 0.2 (1.00)

13. Secondary Outcome: Change From Baseline in EuroQol-5 Dimension-5 Level (EQ-5D-5L) Visual Analog Scale at End of Treatment
Description: The EQ-5D questionnaire is a brief, generic health-related quality of life assessment (HRQOL) that can also be used to incorporate participant preferences into health economic evaluations. The EQ-5D questionnaire assesses HRQOL in terms of degree of limitation on 5 health dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and as overall health using a visual analog scale with response options ranging from 0 (worst imaginable health) to 100 (best imaginable health).
Time Frame: Baseline to EOT (up to 2 years)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ibrutinib+BR | Placebo+BR
Number analyzed (Participants) | 38 | 110
Units on a scale | -4.3 (19.58) | 4.0 (18.21)

14. Secondary Outcome: Change From Baseline in EuroQol-5 Dimension-5 Level (EQ-5D-5L) Utility Score Scale at End of Treatment
Description: The EuroQol-5 is a five dimensional health state classification. Each dimension is assessed on a 3-point ordinal scale (1=no problems, 2=some problems, 3=extreme problems). The responses to the five EQ-5D dimensions were scored using a utility-weighted algorithm to derive an EQ-5D health status index score between 0 to 1. High score indicating a high level of utility.
Time Frame: Baseline to EOT (up to 2 years)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ibrutinib+BR | Placebo+BR
Number analyzed (Participants) | 38 | 110
Units on a scale | 0.0 (0.28) | 0.0 (0.24)

ADVERSE EVENTS:
Time Frame: From the time a signed and dated informed consent form is obtained until 30 days following the last dose of study treatment or until the start of a subsequent systemic antineoplastic therapy, if earlier (up to 5 years)
Description: Safety analysis set included all the randomized participants who received at least 1 dose of study drug or placebo.
Arm/Group | Ibrutinib+BR | Placebo+BR | Crossover to Ibrutinib
All-Cause Mortality (participants affected / at risk) | 74/287 | 107/287 | 57/183
Serious Adverse Events (participants affected / at risk) | 198/287 | 127/287 | 105/183
Other Adverse Events (participants affected / at risk) | 268/287 | 271/287 | 157/183
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrutinib+BR (N=287) | Placebo+BR (N=287) | Crossover to Ibrutinib (N=183)
Anaemia (Blood and lymphatic system disorders) | 3 | 7 | 2
Aplasia Pure Red Cell (Blood and lymphatic system disorders) | 1 | 0 | 0
Aplastic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Autoimmune Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 | 5 | 0
Bone Marrow Failure (Blood and lymphatic system disorders) | 1 | 0 | 0
Cytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 30 | 22 | 2
Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Immune Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 7 | 6 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 2 | 0
Acute Coronary Syndrome (Cardiac disorders) | 0 | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 3 | 1
Angina Pectoris (Cardiac disorders) | 4 | 1 | 0
Angina Unstable (Cardiac disorders) | 1 | 0 | 1
Arrhythmia Supraventricular (Cardiac disorders) | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 16 | 2 | 6
Atrial Flutter (Cardiac disorders) | 1 | 0 | 1
Atrioventricular Block (Cardiac disorders) | 1 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 2 | 0 | 3
Cardiac Failure (Cardiac disorders) | 3 | 0 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 1 | 0 | 0
Cardiopulmonary Failure (Cardiac disorders) | 1 | 0 | 1
Cardiovascular Insufficiency (Cardiac disorders) | 1 | 0 | 0
Carditis (Cardiac disorders) | 1 | 0 | 0
Coronary Artery Occlusion (Cardiac disorders) | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 2 | 2 | 2
Myocarditis (Cardiac disorders) | 1 | 0 | 0
Pericardial Effusion (Cardiac disorders) | 2 | 1 | 1
Sinus Node Dysfunction (Cardiac disorders) | 1 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Ventricular Fibrillation (Cardiac disorders) | 1 | 0 | 0
Ventricular Flutter (Cardiac disorders) | 1 | 0 | 0
Ventricular Tachycardia (Cardiac disorders) | 1 | 0 | 0
Addison's Disease (Endocrine disorders) | 0 | 0 | 1
Goitre (Endocrine disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 3 | 0 | 2
Maculopathy (Eye disorders) | 1 | 0 | 0
Retinal Haemorrhage (Eye disorders) | 0 | 0 | 1
Scleral Disorder (Eye disorders) | 0 | 1 | 0
Vitreous Adhesions (Eye disorders) | 1 | 0 | 0
Vitreous Haemorrhage (Eye disorders) | 1 | 0 | 0
Abdominal Hernia (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal Incarcerated Hernia (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 3
Anal Fistula (Gastrointestinal disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 2 | 0
Colitis Ischaemic (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 0
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Gastric Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Gastric Ulcer Perforation (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 3 | 0 | 0
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Gastrointestinal Inflammation (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 4 | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Intra-Abdominal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Large Intestine Perforation (Gastrointestinal disorders) | 1 | 0 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Mouth Ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal Ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1
Volvulus (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1
Asthenia (General disorders) | 1 | 0 | 0
Chest Pain (General disorders) | 1 | 0 | 0
Chills (General disorders) | 0 | 1 | 0
Complication Associated with Device (General disorders) | 1 | 0 | 0
Condition Aggravated (General disorders) | 1 | 0 | 0
Death (General disorders) | 2 | 0 | 1
Disease Progression (General disorders) | 1 | 2 | 0
Fatigue (General disorders) | 3 | 1 | 1
General Physical Health Deterioration (General disorders) | 1 | 0 | 0
Hernia (General disorders) | 1 | 0 | 0
Influenza Like Illness (General disorders) | 1 | 0 | 0
Infusion Site Extravasation (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 1 | 1 | 1
Mucosal Inflammation (General disorders) | 1 | 1 | 0
Multiple Organ Dysfunction Syndrome (General disorders) | 1 | 3 | 3
Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 0
Oedema Peripheral (General disorders) | 1 | 0 | 0
Pneumatosis (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 11 | 7 | 4
Sudden Cardiac Death (General disorders) | 1 | 0 | 0
Sudden Death (General disorders) | 1 | 0 | 0
Systemic Inflammatory Response Syndrome (General disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis Chronic (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 0
Gallbladder Obstruction (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic Cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis Toxic (Hepatobiliary disorders) | 0 | 2 | 0
Hepatocellular Injury (Hepatobiliary disorders) | 1 | 1 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 1 | 0 | 0
Anaphylactic Reaction (Immune system disorders) | 0 | 1 | 0
Abscess Jaw (Infections and infestations) | 1 | 0 | 0
Actinomycotic Pulmonary Infection (Infections and infestations) | 0 | 1 | 0
Acute Sinusitis (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 2
Arthritis Bacterial (Infections and infestations) | 2 | 0 | 0
Ascariasis (Infections and infestations) | 1 | 0 | 0
Atypical Pneumonia (Infections and infestations) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 2 | 0 | 0
Brain Abscess (Infections and infestations) | 2 | 0 | 0
Breast Abscess (Infections and infestations) | 0 | 0 | 1
Breast Cellulitis (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 8 | 5 | 1
Bronchopulmonary Aspergillosis (Infections and infestations) | 1 | 1 | 2
Campylobacter Infection (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 4 | 2 | 1
Cellulitis Staphylococcal (Infections and infestations) | 1 | 0 | 0
Central Nervous System Infection (Infections and infestations) | 1 | 0 | 0
Chronic Sinusitis (Infections and infestations) | 1 | 1 | 0
Clostridium Difficile Colitis (Infections and infestations) | 0 | 1 | 1
Clostridium Difficile Infection (Infections and infestations) | 0 | 0 | 2
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1
Cytomegalovirus Colitis (Infections and infestations) | 0 | 1 | 0
Cytomegalovirus Infection (Infections and infestations) | 1 | 0 | 0
Dacryocystitis (Infections and infestations) | 1 | 0 | 0
Dermo-Hypodermitis (Infections and infestations) | 0 | 0 | 1
Disseminated Cryptococcosis (Infections and infestations) | 1 | 0 | 0
Epstein-Barr Virus Infection (Infections and infestations) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0 | 3
Escherichia Sepsis (Infections and infestations) | 0 | 0 | 1
Escherichia Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0
Fungal Infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 2 | 0 | 1
Gastrointestinal Infection (Infections and infestations) | 1 | 0 | 0
Haemophilus Infection (Infections and infestations) | 0 | 0 | 1
Hepatitis B Reactivation (Infections and infestations) | 1 | 1 | 0
Herpes Zoster (Infections and infestations) | 1 | 2 | 1
Infection (Infections and infestations) | 3 | 2 | 0
Infectious Pleural Effusion (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 2 | 2
Lung Infection (Infections and infestations) | 3 | 3 | 0
Lymphadenitis Bacterial (Infections and infestations) | 0 | 0 | 1
Muscle Abscess (Infections and infestations) | 0 | 0 | 1
Neutropenic Sepsis (Infections and infestations) | 1 | 0 | 0
Nocardiosis (Infections and infestations) | 1 | 0 | 0
Oral Candidiasis (Infections and infestations) | 0 | 2 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Otitis Media (Infections and infestations) | 1 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 1 | 0
Periorbital Cellulitis (Infections and infestations) | 1 | 0 | 0
Peritonsillar Abscess (Infections and infestations) | 0 | 0 | 1
Pharyngeal Abscess (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Pharyngitis Streptococcal (Infections and infestations) | 1 | 0 | 0
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 2 | 0 | 0
Pneumonia (Infections and infestations) | 48 | 26 | 34
Pneumonia Bacterial (Infections and infestations) | 0 | 1 | 0
Pneumonia Haemophilus (Infections and infestations) | 1 | 0 | 0
Pneumonia Pneumococcal (Infections and infestations) | 1 | 0 | 1
Pneumonia Streptococcal (Infections and infestations) | 0 | 1 | 2
Progressive Multifocal Leukoencephalopathy (Infections and infestations) | 2 | 0 | 2
Pseudomembranous Colitis (Infections and infestations) | 1 | 0 | 0
Pulmonary Tuberculoma (Infections and infestations) | 1 | 0 | 0
Pulmonary Tuberculosis (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Rash Pustular (Infections and infestations) | 1 | 0 | 0
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 5 | 2 | 5
Sepsis (Infections and infestations) | 8 | 4 | 4
Septic Shock (Infections and infestations) | 6 | 2 | 5
Sinusitis (Infections and infestations) | 1 | 2 | 2
Skin Candida (Infections and infestations) | 0 | 0 | 1
Skin Infection (Infections and infestations) | 2 | 1 | 1
Soft Tissue Infection (Infections and infestations) | 1 | 0 | 1
Splenic Abscess (Infections and infestations) | 1 | 0 | 0
Staphylococcal Infection (Infections and infestations) | 2 | 0 | 0
Staphylococcal Skin Infection (Infections and infestations) | 1 | 0 | 0
Subcutaneous Abscess (Infections and infestations) | 3 | 1 | 0
Tooth Abscess (Infections and infestations) | 0 | 1 | 0
Tuberculosis of Central Nervous System (Infections and infestations) | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 3 | 0
Urinary Tract Infection (Infections and infestations) | 6 | 1 | 2
Urosepsis (Infections and infestations) | 1 | 0 | 1
Varicella (Infections and infestations) | 1 | 1 | 0
Varicella Zoster Virus Infection (Infections and infestations) | 0 | 0 | 1
Viral Infection (Infections and infestations) | 0 | 1 | 1
Abdominal Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 2 | 0 | 2
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Incision Site Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 4 | 5 | 0
Pelvic Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pneumoconiosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pneumothorax Traumatic (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 2
Post Procedural Swelling (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Biopsy (Investigations) | 0 | 0 | 1
Blood Creatinine Increased (Investigations) | 1 | 0 | 0
Body Temperature Increased (Investigations) | 0 | 0 | 1
Neutrophil Count Decreased (Investigations) | 2 | 0 | 0
Prostatic Specific Antigen Increased (Investigations) | 0 | 0 | 1
Weight Decreased (Investigations) | 1 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 6 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Chondrocalcinosis Pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Femoroacetabular Impingement (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle Haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Acute Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Adenosquamous Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Anal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1 | 1
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Bronchioloalveolar Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Chronic Myelomonocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Intestinal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Intraductal Papilloma of Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant Melanoma in Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Maxillofacial Sinus Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Myeloproliferative Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neuroendocrine Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal Cancer Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 2
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Superficial Spreading Melanoma Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Carotid Sinus Syndrome (Nervous system disorders) | 1 | 0 | 0
Cerebral Disorder (Nervous system disorders) | 0 | 0 | 1
Cerebral Infarction (Nervous system disorders) | 0 | 0 | 1
Cerebral Ischaemia (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 3 | 0 | 1
Cognitive Disorder (Nervous system disorders) | 1 | 0 | 0
Depressed Level of Consciousness (Nervous system disorders) | 1 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 2
Facial Paresis (Nervous system disorders) | 0 | 1 | 0
Haemorrhage Intracranial (Nervous system disorders) | 1 | 0 | 1
Haemorrhagic Stroke (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Loss of Consciousness (Nervous system disorders) | 0 | 1 | 0
Meningism (Nervous system disorders) | 1 | 0 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 0 | 0
Post Herpetic Neuralgia (Nervous system disorders) | 1 | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 1
Transient Global Amnesia (Nervous system disorders) | 0 | 0 | 1
Vascular Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Acute Stress Disorder (Psychiatric disorders) | 1 | 0 | 0
Alcoholic Psychosis (Psychiatric disorders) | 0 | 0 | 1
Completed Suicide (Psychiatric disorders) | 0 | 1 | 0
Confusional State (Psychiatric disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 1 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 2 | 1 | 0
Calculus Bladder (Renal and urinary disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 2
Nephropathy (Renal and urinary disorders) | 1 | 0 | 0
Nephropathy Toxic (Renal and urinary disorders) | 0 | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0 | 2
Renal Impairment (Renal and urinary disorders) | 2 | 1 | 0
Ureteric Stenosis (Renal and urinary disorders) | 1 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Urge Incontinence (Renal and urinary disorders) | 0 | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 1
Urinary Retention (Renal and urinary disorders) | 1 | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 2 | 0 | 1
Fibrocystic Breast Disease (Reproductive system and breast disorders) | 1 | 0 | 0
Genital Rash (Reproductive system and breast disorders) | 1 | 0 | 0
Pelvic Floor Muscle Weakness (Reproductive system and breast disorders) | 0 | 0 | 1
Penile Dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine Haemorrhage (Reproductive system and breast disorders) | 2 | 0 | 0
Uterine Prolapse (Reproductive system and breast disorders) | 1 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary Sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Respiratory Tract Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute Febrile Neutrophilic Dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Cellulitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Drug Eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Excessive Granulation Tissue (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypersensitivity Vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pemphigus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin Necrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Aortic Aneurysm Rupture (Vascular disorders) | 1 | 0 | 0
Arterial Stenosis (Vascular disorders) | 0 | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 3 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 1
Hypertensive Crisis (Vascular disorders) | 2 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0
Jugular Vein Thrombosis (Vascular disorders) | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 0
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 | 0 | 0
Peripheral Artery Occlusion (Vascular disorders) | 1 | 0 | 0
Peripheral Artery Thrombosis (Vascular disorders) | 1 | 0 | 0
Peripheral Ischaemia (Vascular disorders) | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrutinib+BR (N=287) | Placebo+BR (N=287) | Crossover to Ibrutinib (N=183)
Anaemia (Blood and lymphatic system disorders) | 73 | 79 | 33
Leukopenia (Blood and lymphatic system disorders) | 15 | 18 | 2
Neutropenia (Blood and lymphatic system disorders) | 170 | 159 | 40
Thrombocytopenia (Blood and lymphatic system disorders) | 90 | 69 | 24
Atrial Fibrillation (Cardiac disorders) | 23 | 5 | 19
Cataract (Eye disorders) | 20 | 3 | 8
Dry Eye (Eye disorders) | 15 | 9 | 6
Vision Blurred (Eye disorders) | 19 | 19 | 3
Abdominal Pain (Gastrointestinal disorders) | 39 | 24 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 23 | 16 | 11
Constipation (Gastrointestinal disorders) | 61 | 50 | 15
Diarrhoea (Gastrointestinal disorders) | 115 | 68 | 47
Dyspepsia (Gastrointestinal disorders) | 24 | 21 | 8
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 15 | 12 | 4
Nausea (Gastrointestinal disorders) | 108 | 101 | 16
Toothache (Gastrointestinal disorders) | 15 | 5 | 3
Vomiting (Gastrointestinal disorders) | 42 | 45 | 15
Asthenia (General disorders) | 26 | 24 | 5
Chills (General disorders) | 33 | 31 | 5
Fatigue (General disorders) | 69 | 66 | 32
Influenza Like Illness (General disorders) | 9 | 10 | 12
Mucosal Inflammation (General disorders) | 15 | 7 | 3
Non-Cardiac Chest Pain (General disorders) | 17 | 13 | 3
Oedema Peripheral (General disorders) | 49 | 34 | 21
Pyrexia (General disorders) | 74 | 60 | 22
Bronchitis (Infections and infestations) | 51 | 29 | 19
Cellulitis (Infections and infestations) | 16 | 8 | 10
Conjunctivitis (Infections and infestations) | 20 | 15 | 10
Herpes Zoster (Infections and infestations) | 24 | 17 | 7
Influenza (Infections and infestations) | 22 | 16 | 7
Oral Herpes (Infections and infestations) | 15 | 18 | 7
Pharyngitis (Infections and infestations) | 18 | 13 | 2
Pneumonia (Infections and infestations) | 40 | 25 | 21
Respiratory Tract Infection (Infections and infestations) | 19 | 10 | 15
Sinusitis (Infections and infestations) | 38 | 24 | 25
Upper Respiratory Tract Infection (Infections and infestations) | 69 | 50 | 36
Urinary Tract Infection (Infections and infestations) | 28 | 15 | 26
Contusion (Injury, poisoning and procedural complications) | 30 | 9 | 15
Infusion Related Reaction (Injury, poisoning and procedural complications) | 45 | 64 | 1
Alanine Aminotransferase Increased (Investigations) | 15 | 12 | 3
Blood Creatinine Increased (Investigations) | 17 | 7 | 6
Neutrophil Count Decreased (Investigations) | 21 | 16 | 3
Platelet Count Decreased (Investigations) | 17 | 9 | 2
Weight Decreased (Investigations) | 18 | 18 | 5
Decreased Appetite (Metabolism and nutrition disorders) | 42 | 42 | 16
Hyperuricaemia (Metabolism and nutrition disorders) | 36 | 20 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 24 | 12 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 47 | 29 | 25
Back Pain (Musculoskeletal and connective tissue disorders) | 41 | 22 | 23
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 44 | 14 | 17
Myalgia (Musculoskeletal and connective tissue disorders) | 28 | 15 | 9
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 21 | 15 | 12
Dysgeusia (Nervous system disorders) | 15 | 15 | 3
Headache (Nervous system disorders) | 49 | 47 | 18
Anxiety (Psychiatric disorders) | 22 | 11 | 9
Depression (Psychiatric disorders) | 18 | 8 | 4
Insomnia (Psychiatric disorders) | 27 | 21 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 74 | 75 | 27
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 29 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 22 | 10 | 15
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 16 | 9 | 4
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 30 | 20 | 8
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 18 | 9
Viral Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 30 | 20 | 13
Dry Skin (Skin and subcutaneous tissue disorders) | 27 | 17 | 7
Ecchymosis (Skin and subcutaneous tissue disorders) | 14 | 2 | 10
Onychoclasis (Skin and subcutaneous tissue disorders) | 10 | 0 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 34 | 33 | 9
Rash (Skin and subcutaneous tissue disorders) | 63 | 35 | 15
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 17 | 11 | 7
Skin Lesion (Skin and subcutaneous tissue disorders) | 30 | 5 | 11
Haematoma (Vascular disorders) | 26 | 3 | 14
Hypertension (Vascular disorders) | 47 | 14 | 27

LIMITATIONS AND CAVEATS:
Study was planned to end when 80% of randomized participants died or 5 years after last participant randomized, whichever was first. Sponsor terminated study on 23-Jan-2019 (5 year after last participant randomized) and study was considered completed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT01611090/Prot_000.pdf
  • Statistical Analysis Plan (2015-02-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT01611090/SAP_001.pdf